CLINICAL TRIAL: NCT02728401
Title: Genotypes and Phenotypes in Pediatric SIRS and Sepsis (GAPPSS)
Brief Title: Genotypes and Phenotypes in Pediatric SIRS and Sepsis
Acronym: GAPPSS
Status: Completed | Type: Observational
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Immunexpress (Industry)
Responsible Party: Principal Investigator, Jerry Zimmerman, Professor of Pediatrics and Anesthesiology, Faculty in Pediatric Critical Care Medicine, University of Washington School of Medicine, Seattle Children's Hospital
Other Study IDs: 14761
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Systemic Inflammatory Response Syndrome (SIRS); Sepsis
Keywords: inflammation; sepsis; pediatric; transcripts; serum proteins; cardiopulmonary bypass
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Sepsis; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Type 1: whole blood (2.5 mL) collected daily into PAXgene Blood RNA tube (PreAnalytiX, Ref # 7621650). Type 2: whole blood (1 mL) collected daily into serum separation tube (BD Vacutainer SST™ Tube with Silica Clot Activator, Polymer Gel, Silicone-Coated Interior, Ref # 367983). Type 3: whole blood (1 mL) collected on day 1 into lavender top Vacutainer (BD Vacutainer, lavender top, K2 EDTA 7.2mg, Ref # 367861).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- INSI: Infection-negative systemic inflammation (INSI). The INSI group consists of children who have undergone congenital cardiac defect corrective surgery requiring cardiopulmonary bypass, known to induce an INSI response for ~24 hours thereafter; all children in this cohort are culture negative. This group is demarcated further by inclusion & exclusion criteria (see Eligibility section below).
- CSSS: Clinical severe sepsis syndrome (CSSS). Children assigned to the CSSS group had confirmed or highly suspected infection (microbial culture orders, antimicrobial prescription), exhibited 2 or more systemic inflammatory response syndrome criteria (including temperature and leukocyte criteria), and demonstrated at least cardiovascular ± pulmonary organ dysfunction. This group is demarcated further by inclusion & exclusion criteria (see Eligibility section below).
- Viral: The Viral Infection group consists of children who displayed signs and symptoms of severe viral infection, and who tested positive for respiratory viral infection(s) by a molecular virus panel test. These children were clinically evaluated to not have bacterial sepsis. This group is demarcated further by inclusion & exclusion criteria (see Eligibility section below).

SUMMARY:
The aim of this investigation is to longitudinally quantify host gene expression and serum proteins in children with infectious and non-infectious SIRS. The investigators hypothesize that children with non-infectious SIRS, with bacterial infection associated SIRS, or with viral infection associated SIRS will exhibit distinct patterns of host gene expression and serum proteins. The investigators further hypothesize that it should be possible to discover sets of mRNA or protein biomarkers that will permit unambiguous diagnosis of non-infectious SIRS, SIRS associated with bacterial infection, and SIRS associated with viral infection.

DETAILED DESCRIPTION:
The investigators will undertake a proof-of-concept, pilot, prospective, observational trial that aims to recruit ~90 children from the Seattle Children's Hospital Pediatric Intensive Care Unit (PICU) and Cardiac Intensive Care Unit (CICU). The study will plan to recruit 30 children who are scheduled for surgery to repair congenital cardiac malformations, 15 - 25 immunocompetent children with culture positive sepsis, and 15 - 25 immunocompromised children with culture positive sepsis, and 30-40 children who are polymerase chain reaction (PCR) positive for viral respiratory pathogens (RSV, influenza, parainfluenza, rhinovirus, etc), and who meet the eligibility criteria. In total, accounting for culture negative bacterial sepsis (estimated 40%), the investigators plan to enroll 50 children with sepsis, 30-40 with viral sepsis, and 20 children undergoing surgery for congenital heart disease.

Demographic data will be collected at the time of ICU admission. Illness severity will be quantified by PRISM III and day 1 PELOD scores. Additional measures of sepsis severity will include oxygenation index, saturation index and duration of mechanical ventilation, vasoactive inotropic score and duration of vasoactive-inotropic support and highest serum creatinine on day 1. Resource utilization will be measured as PICU and hospital duration of stay.

For all children enrolled in the study, blood samples will be obtained on study days 1, 2 and 3. For children with sepsis, if cultures remain sterile or PCR negative, no additional research blood samples will be obtained. For children with sepsis and a positive culture or positive PCR by study day 3, additional blood samples will be obtained on the day of PICU discharge.

ELIGIBILITY:
A. INSI group: systemic inflammation, in the absence of culture positive infection. Cardiac surgery patients, n=30.

Inclusion Criteria:

* Admission to the CICU AND
* Age ~1-18 years AND
* Weight exceeding 10 kg
* Vascular catheter capable of providing the blood draw or anticipated orders for venipuncture for clinical labs AND
* Status post open heart surgery requiring cardiopulmonary bypass AND
* Parents speak English AND
* Not previously enrolled in the GAPPSS investigation

Exclusion Criteria:

* Pre- or post-operative culture positive infection OR
* Not expected to survive the CICU stay OR
* Ward of the state OR
* Concurrent malignancy or autoimmune disorder

B. CSSS (Clinical Severe Sepsis Syndrome) group: systemic inflammation, in the presence of highly suspected or documented bacterial infection. Children with clinical severe sepsis, n = 40. In this group, the investigators will enroll children who are immunocompetent as well as children who are immunocompromised.

Inclusion Criteria:

* Admitted to the PICU AND
* Age newborn (>38 weeks EGA)-18 years AND
* Weight equal to or greater than 4 kg AND
* Vascular catheter capable of providing the blood draw or anticipated orders for venipuncture for clinical labs AND
* At least one organ dysfunction (severe sepsis) AND
* Parents speak English AND
* SIRS (systemic inflammatory response syndrome) AND
* Strongly suspected or documented source of infection
* Not previously enrolled in the GAPPSS investigation

Exclusion Criteria:

* PICU nosocomial primary infection accounting for the sepsis event
* Not expected to survive the PICU stay
* Ward of the state

C. Viral Infection group. Severe respiratory dysfunction in the presence of PCR -documented viral infection. Children with clinical severe viral sepsis, n=6. In this group, the investigators will enroll children who are immunocompetent as well as children who are immunocompromised.

Inclusion Criteria:

* Admitted to the PICU AND
* Age newborn (>38 weeks EGA)-18 years AND
* Weight equal to or greater than 4 kg AND
* Vascular catheter capable of providing the blood draw or anticipated orders for venipuncture for clinical labs AND
* Parents speak English AND
* Severe respiratory dysfunction requiring invasive or non-invasive positive pressure mechanical ventilation support AND
* Positive PCR verifying a viral infection
* Not previously enrolled in the GAPPSS investigation

Exclusion Criteria:

* PICU nosocomial primary infection accounting for the sepsis event
* Not expected to survive the PICU stay
* Ward of the state

Ages: 38 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: INSI group: children who had congenital cardiac defect corrective surgery requiring cardiopulmonary bypass, known to induce an INSI response for ~24 hours thereafter. All children in this group were immune competent and culture negative.
  CSSS group: children with confirmed or highly suspected infection (microbial culture orders, antimicrobial prescription), SIRS criteria (including fever/hypothermia and leukocytosis/leukopenia), and at least cardiovascular ± pulmonary organ dysfunction.
  Viral Infection group: children with severe respiratory dysfunction in the presence of PCR -documented viral infection.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Gene Expression Levels | Day 1 of admission to the pediatric intensive care unit (PICU)
  Gene expression levels (quantitative) will be compared between CSSS, INSI and viral infection groups, in a search for signatures that can discriminate these groups

SECONDARY OUTCOMES:
Serum Protein Expression Profiles | Day 1 of admission to the pediatric intensive care unit (PICU)
  Serum protein expression profiles (semi-quantitative) will be compared between CSSS and INSI groups, in a search for signatures that can discriminate the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Jerry J Zimmerman, MD, PhD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to publish the results of the GAPPSS study in a peer-reviewed scientific journal. A supplemental digital file associated with this paper will be made publicly available through a web link, and will contain relevant clinical data (with all patients de-identified).

REFERENCES:
- [Background] Mathias B, Mira JC, Larson SD. Pediatric sepsis. Curr Opin Pediatr. 2016 Jun;28(3):380-7. doi: 10.1097/MOP.0000000000000337. PMID 26983000
- [Background] Weiss SL, Fitzgerald JC, Pappachan J, Wheeler D, Jaramillo-Bustamante JC, Salloo A, Singhi SC, Erickson S, Roy JA, Bush JL, Nadkarni VM, Thomas NJ; Sepsis Prevalence, Outcomes, and Therapies (SPROUT) Study Investigators and Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. Global epidemiology of pediatric severe sepsis: the sepsis prevalence, outcomes, and therapies study. Am J Respir Crit Care Med. 2015 May 15;191(10):1147-57. doi: 10.1164/rccm.201412-2323OC. PMID 25734408
- [Result] Zimmerman JJ, Sullivan E, Yager TD, Cheng C, Permut L, Cermelli S, McHugh L, Sampson D, Seldon T, Brandon RB, Brandon RA. Diagnostic Accuracy of a Host Gene Expression Signature That Discriminates Clinical Severe Sepsis Syndrome and Infection-Negative Systemic Inflammation Among Critically Ill Children. Crit Care Med. 2017 Apr;45(4):e418-e425. doi: 10.1097/CCM.0000000000002100. PMID 27655322
- [Result] McHugh L, Seldon TA, Brandon RA, Kirk JT, Rapisarda A, Sutherland AJ, Presneill JJ, Venter DJ, Lipman J, Thomas MR, Klein Klouwenberg PM, van Vught L, Scicluna B, Bonten M, Cremer OL, Schultz MJ, van der Poll T, Yager TD, Brandon RB. A Molecular Host Response Assay to Discriminate Between Sepsis and Infection-Negative Systemic Inflammation in Critically Ill Patients: Discovery and Validation in Independent Cohorts. PLoS Med. 2015 Dec 8;12(12):e1001916. doi: 10.1371/journal.pmed.1001916. eCollection 2015 Dec. PMID 26645559